CLINICAL TRIAL: NCT01360164
Title: Phase I/II Study of Umbilical Cord Mesenchymal Stem Cell Therapy for Patients With Hereditary Ataxia
Brief Title: Safety and Efficacy of Umbilical Cord Mesenchymal Stem Cell Therapy for Patients With Hereditary Ataxia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Beike Bio-Technology Co., Ltd. (Industry)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Nanjing Medical University (Other); Nanjing University Medical College Affiliated Wuxi Second Hospital (Unknown); Xuzhou Medical University (Other); The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BKCR-HA-1.0(2010)
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Hereditary Ataxia
Keywords: Human Umbilical Cord Mesenchymal Stem Cells
MeSH Terms: conditions — Spinocerebellar Degenerations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Human umbilical cord mesenchymal stem cells transplantation (Experimental): Participants will be given umbilical cord mesenchymal stem cells transplantation with a 1 year follow-up.
  Interventions: Biological: human umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: human umbilical cord mesenchymal stem cells — Participants will be given hUC-MSCs transplantation.
  Other Names: Intervention Group

SUMMARY:
The Hereditary Ataxias are a group of genetic disorders characterized by slowly progressive incoordination of gait and often associated with poor coordination of hands, speech, and eye movements. Current treatments for Hereditary Ataxias are mainly pharmacological, rehabilitative, or psychological treatments，while no effective treatment available. Stem Cell therapy is a novel and promising therapeutic strategy for Hereditary Ataxias treatment. In this study, the safety and efficacy of Human Umbilical Cord Mesenchymal Stem Cells transplantation will be evaluated in patients with Hereditary Ataxias.

DETAILED DESCRIPTION:
This Study is designed to evaluate the the safety and efficacy of Human Umbilical Cord Mesenchymal Stem Cells transplantation in patients with Hereditary Ataxias.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16-65 years.
* Harding Diagnosis of SCAs, gene type confirmed.
* Candidates who did not receive any stem cell therapy in past 6months.
* sign the consent form and follow the clinic trail procedure.

Exclusion Criteria:

* Cardiac insufficiency; Renal insufficiency; hepatic insufficiency; Total bilirubin higher than 1.5 times of upper limit of normal value; AST /ALT higher than 2.5 times of upper limit of normal value；
* Routine Blood Test: WBC count <3.0×109/ L; PLT count <5×109/L ; or Hemoglobin <100g/L；
* Combined Pneumonia or other Severe systemic bacteria infection；
* Severe drug allergic history or anaphylaxis to 2 or more food or medicine；
* Other brain organic disease (eg. Brain cancer)；
* HIV+, Tumor Markers + ；
* Severe psychotic patients, cognitive dysfunction， or can not understand or sign the Consent Form；
* Other severe systemic or organic disease；
* Uncontrolled hypertension，blood pressure≥180mmHg/110 mmHg after treatment；
* Pregnancy；
* Enrollment in other trials in the last 3 months；
* Other criteria the investigator consider improper for inclusion.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
scores of International Cooperative Ataxia Rating Scale （ICARS） scale and Berg Scale | 1 year after treatment
the volume of Cerebellum of Brain Magnetic Resonance Imaging （MRI） Scan | 1 year after treatment

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 1 year after treatment
Number of Participants with Serious Adverse Events as a Measure of Safety and Tolerability | 1 year after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing University Medical College Affiliated Drum Tower Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Jin JL, Liu Z, Lu ZJ, Guan DN, Wang C, Chen ZB, Zhang J, Zhang WY, Wu JY, Xu Y. Safety and efficacy of umbilical cord mesenchymal stem cell therapy in hereditary spinocerebellar ataxia. Curr Neurovasc Res. 2013 Feb;10(1):11-20. doi: 10.2174/156720213804805936. PMID 23151076